CLINICAL TRIAL: NCT03020927
Title: Therapist and Parent Delivered Reciprocal Imitation Training for Young Children With Autism Spectrum Disorder
Acronym: ParentRIT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently do not have resources/staff to enroll new participants.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Katherine Walton, Assistant Professor of Psychology and Psychiatry, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015B0475
Record Dates: First submitted 2016-06-03; First posted 2017-01-13 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapist Delivered (Active Comparator): Children in the therapist-delivered condition will receive two, 60-minute long sessions of Reciprocal Imitation Training each week for ten consecutive weeks. These sessions will be delivered by trained graduate, undergraduate, and post-graduate research staff. Parents will be permitted to observe sessions via live video, but will not be directly involved in intervention.
  Interventions: Behavioral: Reciprocal Imitation Training (Therapist-Delivered)
- Parent + Therapist Delivered (Experimental): Children in the parent + therapist-delivered condition will receive one, 60-minute long session of Reciprocal Imitation Training each week for ten consecutive weeks. These sessions will be delivered by trained graduate, undergraduate, and post-graduate research staff. During the same period of time, parents/guardians of children will receive one, 60-minute long parent education session per week with graduate and post-graduate research staff, aimed at teaching parents to implement Reciprocal Imitation Training at home with the child.
  Interventions: Behavioral: Reciprocal Imitation Training (Therapist + Parent Delivered)

INTERVENTIONS:
Behavioral: Reciprocal Imitation Training (Therapist-Delivered) — Naturalistic Developmental Behavioral Intervention aimed at improving social imitation skills.
  Other Names: RIT
  Arms: Therapist Delivered
Behavioral: Reciprocal Imitation Training (Therapist + Parent Delivered) — Naturalistic Developmental Behavioral Intervention aimed at improving social imitation skills, using a combination of therapist-delivered intervention and parent training to deliver intervention in the home setting.
  Other Names: RIT
  Arms: Parent + Therapist Delivered

SUMMARY:
The purpose of this study is to examine whether adding a parent education component to an existing intervention (Reciprocal Imitation Training) results in improved outcomes for children with Autism Spectrum Disorder. Reciprocal Imitation Training (RIT) is a behavioral intervention designed to improve spontaneous imitation skills in young children with Autism Spectrum Disorder (ASD). Previous research suggests that it can be effective when used by trained therapists, teachers, siblings, and parents of children with ASD. However, it is unclear to what extent training parents to use RIT strategies in the home environment may enhance outcomes, compared to having therapists implement RIT individually with the child. The study will compare two different versions of RIT for young children with ASD: (1) two 60-minute weekly sessions of therapist-implemented RIT and (2) one weekly 60-minute session of therapist-implemented RIT and one weekly 60-minute session of parent education about using RIT in the home environment. The investigators will examine child and family outcomes between these two intervention types. Outcomes examined will include: (1) spontaneous and prompted imitation skills in the child with ASD, (2) social communication skills in the child with ASD, (3) parent stress, and (4) parent and child behaviors during parent-child play interactions.

ELIGIBILITY:
Inclusion Criteria:

* have a community diagnosis of Autism Spectrum Disorder (as reported by parent)
* meet cutoff for "Autism" or "Autism Spectrum" on the Autism Diagnostic Observation Schedule, 2nd Edition
* be between 24 and 60 months of age at the time of study enrollment
* demonstrate difficulties with imitation skills on the Motor Imitation Scales and/or the Unstructured Imitation Assessment during pre-treatment assessments

Exclusion Criteria:

* Participants must not be the sibling of another study participant

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Unstructured Imitation Assessment (UIA) | Change from baseline to 10 weeks (immediately post-intervention)
  The Unstructured Imitation Assessment (UIA) is a semi-structured, standardized test of imitation skills containing 10 object imitation and 10 gesture imitation tasks (Ingersoll & Meyer, 2011).
Percentage of parent acts imitated during Parent-Child Play Interaction | Change from baseline to 10 weeks (immediately post-intervention)
  Percentage of parent play acts and meaningful gestures imitated by the child during a 10-minute unstructured play interaction with parent

SECONDARY OUTCOMES:
Parenting Stress Index, 4th Edition | Change from baseline to 10 weeks (immediately post-intervention)
Motor Imitation Scales | 10 weeks (immediately post-intervention), 3 months post-treatment, 6 months post-treatment
Early Social Communication Scales | 10 weeks (immediately post-intervention), 3 months post-treatment, 6 months post-treatment
Proportion of time spent jointly engaged during Parent-Child Play Interaction | Change from baseline to 10 weeks (immediately post-intervention)
  Proportion of time spent in joint engagement state (joint focus on same activity) during a 10-minute unstructured play interaction with parent

OTHER OUTCOMES:
Modified Behavior Intervention Rating Scale | 10 weeks (immediately post-intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No